CLINICAL TRIAL: NCT06929585
Title: Genicular Artery Embolization (GAE) vs inTra-articular Corticosteroid Injection for Osteoarthritic Knee Pain. (GET-IN Study)
Brief Title: Genicular Artery Embolization (GAE) vs inTra-articular Corticosteroid Injection for Osteoarthritic Knee Pain.
Acronym: GET-IN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was terminated due to infeasible enrollment. Only one participant was enrolled, and the comparator arm was not initiated.
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202408153RIND
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: knee osteoarthritis; genicular artery embolization; imipenem/cilastatin; intra-articular corticosteroid injection
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: GAE (IPM/CS). (Experimental): Genicular artery embolization with imipenem/cilastatin (IPM/CS).
  Interventions: Procedure: Genicular artery embolization
- Comparator: IA (corticosteroids) (Active Comparator): The patient will receive IA procedure and sham GAE procedure.
  Interventions: Procedure: Intra-articular injection with corticosteroids.

INTERVENTIONS:
Procedure: Genicular artery embolization — The patient will receive GAE procedure and sham IA procedure.
  Arms: Experimental arm: GAE (IPM/CS).
Procedure: Intra-articular injection with corticosteroids. — The patient will receive IA procedure and sham GAE procedure.
  Arms: Comparator: IA (corticosteroids)

SUMMARY:
This study investigates genicular artery embolization (GAE) as a minimally invasive alternative to ntra-articular corticosteroid injections (IA) or treating knee osteoarthritis (OA) pain. Designed as a randomized controlled tria, the study compares pain relief effectiveness and safety between GAE and IA over a 12-month follow-up. Eligible participants are aged over 40 with symptomatic knee OA resistant to conservative treatment. Primary outcomes focus on pain reduction (NRS score), while secondary measures include function, quality of life, imaging findings, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Symptomatic knee pain, with numeric rating scale (NRS) ≥ 4.
3. Insufficient or resistant to conservative treatment, including oral analgesics, physical therapy, intra-articular injections for at least 3 months, before the enrollment.
4. Weight bearing X ray of knee: osteoarthritis of Kellgren-Lawrence grade 1, 2, or 3.

Exclusion Criteria:

1. History of trauma in recent 6 months.
2. Bleeding tendency.
3. Poor renal function (serum creatinine > 2.0 mg/dL).
4. Pregnancy or breast-feeding.
5. Severe peripheral arterial occlusive disease (PAOD).
6. Local infections or inflammatory arthritis of knee.
7. Rheumatoid arthritis or other rheumatological diseases.
8. Prior knee surgeries (arthroscopic surgery, menisci repair, cruciate ligament reconstruction, arthroplasty of knee) due to knee pain.
9. Malignancy
10. ECOG > grade 2
11. Life expectancy less than 2 years.
12. Any other condition related to the patient's health, regarded exclusionary in the opinion of the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: numeric rating scale (NRS) | Post-intervention 3 month.
  Changes of pain score (NRS) at the 3-month compared with the baseline.

SECONDARY OUTCOMES:
Clinical Efficacy: numeric rating scale (NRS) | In the one-year period after intervention.
  Maximum decreased of pain score (NRS)
Clinical Efficacy: WOMAC | Pre-intervention, post-1, 3, 6, 12 months
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
  *Clinical success defined as ≥ 40% improvement of the WOMAC score.
Clinical Efficacy: Lequesne'Index | Pre-intervention, post-1, 3, 6, 12 months
  Lequesne index for knee osteoarthritis severity.
Clinical Outcome: PGIC | Pre-intervention, post-1, 3, 6, 12 months
  Self-report measure Patient Global Impression of Change (PGIC).
Clinical Outcome: Analgesic Usage and other Pain Control Treatments | Pre-intervention, post-1, 3, 6, 12 months
  Use of narcotics or non-steroidal anti-inflammatory drugs (NSAID's); other pain control treatments.
Clinical Outcome: Quality of Life | Pre-intervention, post-1, 3, 6, 12 months
  EQ-5D-5L questionnaire

OTHER OUTCOMES:
Adverse Events Monitoring | Pre-intervention, post-1, 3, 6, 12 months
  The society of interventional radiology AE classification system, 2017 modification.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hosiptal Yunlin Branch, Douliu, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: No